CLINICAL TRIAL: NCT02314884
Title: A Phase I, Open-label, Dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of Cafusertib Hydrochloride in Patients With Advanced Solid Tumors
Brief Title: Phase I Trial to Investigate Cafusertib Hydrochloride Monotherapy in Chinese Patients With Advanced Solid Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10159-I-02
Record Dates: First submitted 2014-12-08; First posted 2014-12-11 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cafusertib Hydrochloride (Experimental): Cafusertib Hydrochloride d1q3w
  Interventions: Drug: Cafusertib Hydrochloride

INTERVENTIONS:
Drug: Cafusertib Hydrochloride

SUMMARY:
A Phase I, Open-label, Dose-escalation Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumor Activity of Cafusertib Hydrochloride in Patients With Advanced Solid Tumors

DETAILED DESCRIPTION:
To investigate safety, tolerability of cafusertib in Chinese patients with Advanced Solid Tumors that are not eligible for conventional or intensive treatment. The dose of cafusertib will be escalated to determine the dose limiting toxicity (DLT) and the maximum tolerated dose (MTD) of cafusertib in advanced cancer patients. At the same time, pharmacokinetic characteristics and preliminary efficacy of cafusertib will be observed in advanced cancer patients. To determine the recommended dosage regimen for phase II.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients age 18 years to 75 years at the time of informed consent
* Eastern Cooperative Oncology Group performance status score of 0-2 at screening
* Life expectancy of at least 12 weeks
* At least one target tumor lesion has not been irradiated and can accurately be measure.

Patients with histologically or cytologically confirmed diagnosis of advanced solid tumors, who had failed conventional treatment, or for whom no therapy of efficacy existed.

Signed informed consent consistent with Chinese Good Clinical Practice.

Male or female patients of child-producing potential must agree to use appropriate contraceptive measures (hormones or barrier or abstinence) during the study and for 90 days after the last day of treatment, serum pregnancy test must be negative within 7 days prior to initiation of study treatment, infertile women is defined as hysterectomy, ovariotomy or menopause for at least 12 months.

Adequate bone marrow, renal and hepatic function parameters: ANC more than 2000/mm3, platelet count more than 100 000/mm3, hemoglobin more than 90 g/L; Total bilirubin less than 1.5 x upper limit of normal，ALT and AST less than 2.5 x upper limit of normal，less than 5.0 x upper limit of normal in case of liver metastases; serum creatinine less than 1.5 x upper limit of normal, creatinine clearance rate more than 50 ml/min (as calculated according to Cockcroft-Gault formula for GFR estimate); Relatively normal ECG (electrocardiogram), QT intervals below 450 ms (male) ,QT intervals below 470 ms (female); LVEF more than 50%.

Exclusion Criteria:

Uncontrolled accumulation of coelomic fluid.

Any anti-cancer therapy, including chemotherapy, hormonal therapy, biologic therapy or radiotherapy within 4 weeks prior to initiation of study treatment, or received nitrourea or mitomycin chemotherapy within 6 weeks prior to initiation of study treatment.

* Side effects/toxicities of such surgery that have not recovered to CTCAE grade 1
* Patients who can't be interrupted use drugs, which may cause QT prolongation (see annex 2)
* Patients with meningioma or current symptomatic brain metastases
* Co-existing malignancy or malignancies diagnosed within the last 5 years with the exception of completely removed skin basal cell carcinoma or cervical cancer in situ
* Concurrent anti-tumor therapy
* Involved in other clinical trials less than 4 weeks prior to Day 1
* Known hypersensitivity to more than two substances or the trial drugs and their excipients
* Patients with serious infections
* Patients with history of immune deficiency, including positivity to HIV antibody, or other acquired, congenital immunodeficiency disease, or history of organ transplantation
* Known positivity to hepatitis B antigen or hepatitis C antibody
* Patient with other serious diseases, in the investigator's opinion, can bring patients great risk. Including but not limited to the following: unstable cardiac diseases (history of myocardial infarction within 6 months prior to Day 1, New York Heart Association Class III or greater, with poorly controlled atrial fibrillation or hypertension), need long-term steroids or immunosuppressive therapy of diseases, such as rheumatoid arthritis, multiple sclerosis and systemic lupus erythematosus
* Pregnant(positive pregnancy test) or lactating women
* Active alcohol abuse or heavy smoker
* A previous history of neurological or psychiatric disorders, including epilepsy or dementia
* Subject is thought unfit for this study by investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
MTD of cafusertib based on the incidence of dose limiting toxicities | 4 weeks

SECONDARY OUTCOMES:
Objective response rate (ORR) according to Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 | 6 weeks
Incidence and intensity of Adverse Events according to Common Toxicity Criteria for AEs (CTCAE version 4.0) | 6 weeks
Occurrence of dose limiting toxicities (DLT) | 4 weeks
Max concentration (Cmax) of cafusertib | 3 weeks
AUC of cafusertib | 3 weeks
Elimination half-life(T1/2) of cafusertib | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China